CLINICAL TRIAL: NCT06538740
Title: A Randomized Trial Investigating the Impact of High Versus Lower Oxygen Fraction During Extubation on Postoperative Pulmonary Atelectasis Measured With Electrical Impedance Tomography
Brief Title: Impact of High Versus Lower Oxygen Fraction Prior to Extubation on Postoperative Pulmonary Atelectasis Measured With EIT
Acronym: RESPIRA-EIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Maximilian S Schaefer, Director of the Center for Anesthesia Research Excellence (CARE) Division Director of Thoracic Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB: 2023P000223
Record Dates: First submitted 2024-07-02; First posted 2024-08-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Atelectasis
Keywords: Pulmonary Atelectasis [C08.381.730]; Oxygen [D01.268.185.550, D01.362.670]; Electrical impedance tomography; Center of Ventilation; lung aeration; anesthesia
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: This study is a single blinded, randomized, trial comparing two study groups ("intervention" and "control")
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Ventilating the patient with 100% oxygen concentration during the wash out phase, before extubation
- Intervention group (Active Comparator): Ventilating the patient with lower (40 or 70%) oxygen concentration during the wash out phase, before extubation
  Interventions: Procedure: Ventilating the patient with lower (40 or 70%) oxygen concentration during the wash out phase, before extubation

INTERVENTIONS:
Procedure: Ventilating the patient with lower (40 or 70%) oxygen concentration during the wash out phase, before extubation — The investigated intervention is the application of 70% inspired oxygen compared to 100% inspired oxygen during the anesthetic washout, right before extubation of the patient for the first 24 enrolled patients, and 40% inspired oxygen compared to 100% inspired oxygen for the subsequently enrolled 24 patients. Before and after the intervention EIT measurements are performed at designated time points to assess lung aeration and calculate the center of ventilation. This information allows assumptions on atelectasis formation in the patients' lung.
  Arms: Intervention group

SUMMARY:
Patients undergoing general anesthesia require mechanical ventilation (artificial delivery of air and oxygen to their lungs). It is well known that during mechanical ventilation, so-called atelectasis formation occurs. This is a condition characterized by partial or complete collapse of lung tissue that can result in a reduction in oxygen uptake through the lung. A known risk factor for atelectasis formation during mechanical ventilation is the utilization of high oxygen concentration, as the oxygen molecules are absorbed in the lung, which then can lead to collapse of the tissue. Despite the proven association, standard operating procedure at the end of anesthesia still requires utilization of 100% oxygen. Its justification is the goal to ensure sufficient oxygenation throughout the extubation phase. However, clinical observation doesn't show a lack of oxygenation in this phase, but the patient is still exposed to the risk of atelectasis formation.

This study aims to investigate the hypothesis of whether the utilization of reduced inspiratory oxygen concentration before extubation (70% or 40% compared to 100%) reduces atelectasis formation. The study was originally planned to randomize 24 patients to either 70% or 100% inspiratory oxygen concentration at the end of anaesthesia. After completion of this first phase, the study was amended to enroll another 24 patients randomized to 40% or 100% inspiratory oxygen concentration at the end of anaesthesia.

Of note, both concentrations are still higher than when breathing room air in, which has of 21% oxygen. During the intervention, parameters such as the oxygen content in the blood (oxygen saturation, SpO₂), heart rate, and blood pressure are recorded, and atelectasis formation is measured using a technique called electrical impedance tomography (EIT). EIT measurements are performed at designated time points during the procedure. Anesthesia care providers are asked to document procedural, patient, and ventilator data in a questionnaire. Secondary outcomes are the homogeneity and distribution of air measured with EIT, as well as some clinical outcomes including post-extubation desaturation (<90% SpO₂), incidence of re-intubation or non-invasive ventilation, and the Post-anesthesia Care Unit (PACU) length of stay.

DETAILED DESCRIPTION:
This study is a single blinded randomized controlled trial with and aims to assess whether the use of 100% oxygen before extubation favors postoperative atelectasis formation compared to the use of lower oxygen concentrations whilst still ensuring patient safety. The study was originally planned to randomize 24 patients to either 70% or 100% inspiratory oxygen concentration at the end of anaesthesia. After completion of this first phase, the study was amended to enroll another 24 patients randomized to 40% or 100% inspiratory oxygen concentration at the end of anaesthesia. Patients are randomized to either the control group or the intervention group.

The randomization scheme is developed by a non-blinded statistician using the Statistical Analysis Software (SAS) and uploaded to the Research Electronic Data Capture (REDCap) randomization module, enabling delegated team members to generate sequential allocations for enrolled subjects.

Screening of potential study subjects is performed by the PI. The patient is asked to participate in the study by the PI or co-investigator and the study design and procedures are explained to the patient, while they are still in the holding area on the day of the procedure.

The patients in both groups (control and intervention) are equipped with the EIT belt as well as an additional SpO₂ recording device before induction and intubation. After onset of mechanical ventilation as per institutional standards, an inspiratory oxygen concentration of 50% is aimed. Actual oxygen concentration as well as any administration of drugs remain at the discretion of the anesthesia care provider. At the end of the procedure, before the initiation of volatile anesthetic washout, fresh gas flow is increased to 15 liters per minute (or the highest fresh gas flow allowed at the respective anesthesia machine if 15 liters per minute cannot be achieved), and a fraction of inspired oxygen (FiO₂) of either 70% (intervention group) or 100% (control group) for the first 24 randomized patients, and of either 40% (intervention group) or 100% for the subsequent 24 randomized patients is applied.

EIT measurements take place at 6 designated time points before, during and after the procedure. These time points are: Pre-induction, after intubation, just before washout, pre-extubation, one minute after extubation and 60 minutes after extubation in the PACU.

The primary outcome for the study is the Center of Ventilation (CoV), measured through electrical impedance tomography (EIT) compared at one minute after extubation between the control group and intervention groups.

Secondary outcomes include the homogeneity index, and the distribution of lung aeration measured by EIT. In addition, we measure the peripheral oxygen concentration during the whole interventional period and during the PACU stay to evaluate any occurrence of desaturation (SpO₂ <90%) within the first 60 minutes after extubation in the PACU. The incidence of re-intubation or the need for non-invasive ventilation in the next 7 days and an unplanned admission, to either ICU, Intermediate Care Unit (IMC) or the normal ward, as well as the length of stay in the PACU are other clinical secondary outcomes compared between the groups. Subsequent analyses will assess differences between the 70% and 40% oxygen subgroups within the intervention arm to evaluate potential dose-dependency.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Elective surgery with general anesthesia and endotracheal intubation
* Expected duration of surgery 1-5 hours
* Consent obtained from patient

Exclusion Criteria:

* Patients with inability to give written informed consent
* American Society of Anesthesiologists (ASA) physical status> IV
* Morbid obesity BMI > 40
* Suspected pregnancy and lactation
* Cardiac or thoracic surgery
* Patients with thoracic epidural catheters
* Patients with active implantable devices, such as pacemakers, cardioverter defibrillators, or neurostimulators
* Compromised airways
* Impaired oxygenation at baseline or during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
The shift of Center of Ventilation (CoV), measured through Electrical Impedance Tomography (EIT) in %. | The CoV is measured at six points: pre-induction, post-intubation, pre-washout, pre-extubation, 1 min post-extubation, and 60 min post-extubation in the PACU. The primary outcome is the difference between pre-induction and 1 min post-extubation.
  The Center of Ventilation (CoV) is a variable based on the EIT. It is calculated after the initial measurements and defines the most ventilated area of the lung. Assumptions on atelectasis formation can be drawn when the CoV shifts to more ventral areas than measured before. Primary outcome is the absolute difference between the first measurement (before induction) and the measurement directly after extubation in %.

SECONDARY OUTCOMES:
The 1st secondary outcome is the variation of the inhomogeneity index within each patient, measured through Electrical Impedance Tomography (EIT). | The inhomogeneity index is measured at six points: pre-induction, post-intubation, pre-washout, pre-extubation, 1 min post-extubation, and 60 min post-extubation in the PACU.
  The inhomogeneity index is a variable based on the EIT and is calculated after the initial measurements. It defines the homogeneity of the aeration throughout the whole ventilated area and provides information on potential atelectasis formation or overventilation in certain lung areas. The outcome is the variation of the inhomogeneity index within each patient.
The 2nd secondary outcome is the distribution of lung aeration, measured through Electrical Impedance Tomography (EIT). | The distribution of lung aeration is measured at six points: pre-induction, post-intubation, pre-washout, pre-extubation, 1 min post-extubation, and 60 min post-extubation in the PACU.
  The distribution is a variable based on the EIT and can be calculated after the initial measurements. It defines the distribution of the lung aeration throughout the whole ventilated area and can give information on potential atelectasis formation in the lung.
Minutes of hypoxemia in the first 60 minutes after extubation | The SpO2 data analysis starts with the time the patient enters the PACU and is continued until the patient is discharged from the PACU, which is typically one to two hours after the end of surgery.
  It is determined as SpO2 < 90% for more than two minutes throughout the stay in the PACU in the first 60 minutes after extubation.
Re-intubation or the need for unplanned non-invasive ventilation within 7 days. | 7 days post-operative
  It is determined as re-intubation or the need for unplanned non-invasive ventilation (NIV).
Unplanned admission to either ICU, IMC or a normal unit. | Unplanned admission to either ICU, ICM or a normal unit after the PACU stay is determined in the time frame after end of surgery and up to 7 days after the surgery.
  Number of patients that experience unplanned admission to either ICU, IMC or a normal unit after their PACU stay.
Length of stay in the PACU | The length of stay in the PACU is measured in minutes from admission to discharge from the PACU.
  It is determined as the length of stay in the PACU in minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia, Critical Care and Pain Medicine, Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frerichs I, Amato MB, van Kaam AH, Tingay DG, Zhao Z, Grychtol B, Bodenstein M, Gagnon H, Bohm SH, Teschner E, Stenqvist O, Mauri T, Torsani V, Camporota L, Schibler A, Wolf GK, Gommers D, Leonhardt S, Adler A; TREND study group. Chest electrical impedance tomography examination, data analysis, terminology, clinical use and recommendations: consensus statement of the TRanslational EIT developmeNt stuDy group. Thorax. 2017 Jan;72(1):83-93. doi: 10.1136/thoraxjnl-2016-208357. Epub 2016 Sep 5. PMID 27596161
- [Background] Riva T, Pascolo F, Huber M, Theiler L, Greif R, Disma N, Fuchs A, Berger-Estilita J, Riedel T. Evaluation of atelectasis using electrical impedance tomography during procedural deep sedation for MRI in small children: A prospective observational trial. J Clin Anesth. 2022 May;77:110626. doi: 10.1016/j.jclinane.2021.110626. Epub 2021 Dec 10. PMID 34902800
- [Background] Schaefer MS, Wania V, Bastin B, Schmalz U, Kienbaum P, Beiderlinden M, Treschan TA. Electrical impedance tomography during major open upper abdominal surgery: a pilot-study. BMC Anesthesiol. 2014 Jul 5;14:51. doi: 10.1186/1471-2253-14-51. eCollection 2014. PMID 25018668
- [Background] Victorino JA, Borges JB, Okamoto VN, Matos GF, Tucci MR, Caramez MP, Tanaka H, Sipmann FS, Santos DC, Barbas CS, Carvalho CR, Amato MB. Imbalances in regional lung ventilation: a validation study on electrical impedance tomography. Am J Respir Crit Care Med. 2004 Apr 1;169(7):791-800. doi: 10.1164/rccm.200301-133OC. Epub 2003 Dec 23. PMID 14693669
- [Background] Benoit Z, Wicky S, Fischer JF, Frascarolo P, Chapuis C, Spahn DR, Magnusson L. The effect of increased FIO(2) before tracheal extubation on postoperative atelectasis. Anesth Analg. 2002 Dec;95(6):1777-81, table of contents. doi: 10.1097/00000539-200212000-00058. PMID 12456458
- [Background] Rothen HU, Sporre B, Engberg G, Wegenius G, Reber A, Hedenstierna G. Prevention of atelectasis during general anaesthesia. Lancet. 1995 Jun 3;345(8962):1387-91. doi: 10.1016/s0140-6736(95)92595-3. PMID 7760608
- [Background] Reber A, Engberg G, Wegenius G, Hedenstierna G. Lung aeration. The effect of pre-oxygenation and hyperoxygenation during total intravenous anaesthesia. Anaesthesia. 1996 Aug;51(8):733-7. doi: 10.1111/j.1365-2044.1996.tb07885.x. PMID 8795314